CLINICAL TRIAL: NCT06008158
Title: Prospective Evaluation of a Once Per Day Regimen of Accelerated Partial Breast Irradiation in Low-Risk, Hormone-Responsive Breast Cancer
Brief Title: Evaluation of a Once Per Day Regimen of Accelerated Partial Breast Irradiation for Improved Breast Appearance in Pts w/Low Risk, Hormone Responsive Brst Ca
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: accrual goals
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 23037; NCI-2023-05718 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23037 (Other: City of Hope Comprehensive Cancer Center); P30CA033572 (NIH)
Record Dates: First submitted 2023-08-18; First posted 2023-08-23 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Anatomic Stage 0 Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Estrogen Receptor-Positive Breast Carcinoma; HER2-Negative Breast Carcinoma
MeSH Terms: conditions — Breast Carcinoma In Situ

STUDY DESIGN:
Masking Description: Cosmetic outcome assessed by blinded medical doctor review.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Supportive care (APBI) (Experimental): Patients undergo APBI QD on consecutive business days for 5 treatments.
  Interventions: Radiation: Accelerated Partial Breast Irradiation

INTERVENTIONS:
Radiation: Accelerated Partial Breast Irradiation — Undergo APBI
  Other Names: Accelerated Partial Breast Radiation Therapy; APBI

SUMMARY:
This phase II trial tests how well accelerated partial breast irradiation (APBI) delivered once per day works in ensuring an acceptable breast appearance in patients with low risk, hormone responsive breast cancer. APBI uses precise radiation beams to kill cancerous cells in a smaller area of the breast (partial breast) instead of the whole breast or chest area as in standard therapy. Additionally, APBI is given in a shorter course of treatment than whole breast radiation therapy, over fewer days instead of several weeks, with a lower total dose of radiation. APBI is currently given every other business day for a total of 5 treatments with excellent results; however, a shorter treatment duration could have similar or even better results. Undergoing APBI every day on consecutive business days for 5 treatments may result in an improved breast appearance for patients with low risk hormone responsive breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish that APBI delivered once per day (APBI QD) for low-risk breast cancer patients results in acceptable patient-reported cosmetic appearance of the breast at 1 year after completion of APBI QD.

SECONDARY OBJECTIVES:

I. To determine the long-term patient-reported cosmetic appearance of the breast in patients treated with APBI QD.

II. To determine the short-term and long-term physician reported cosmetic appearance of the breast in patients treated with APBI QD.

III. To determine the acute and late patient-reported radiation toxicity of APBI QD.

IV. To determine the acute and late physician-reported radiation toxicity of APBI QD.

V. To determine the cancer control outcomes of APBI QD.

EXPLORATORY OBJECTIVES:

I. To assess the health-related quality of life in patients treated with APBI QD.

II. To determine the long-term blinded physician review of cosmetic appearance of the breast in patients treated with APBI.

III. To assess dosimetric parameters associated with cosmesis in patients undergoing APBI QD.

OUTLINE:

Patients undergo APBI QD on consecutive business days for 5 treatments.

Patients follow up at 1 month, 6 months, and 1 year post-APBI and then yearly until 5 years post-APBI.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative
* Age: >= 40 years
* Female
* Ability to read and understand English or Spanish for questionnaires
* Anatomic pathologic stage 0 (ductal carcinoma in situ [DCIS]) or stage IA (invasive) breast cancer
* Malignancy must be epithelial. Non-epithelial breast malignancies such as lymphoma or sarcoma are not allowed
* Tissue from core biopsy or resection must show hormone sensitive receptors. Hormone sensitive receptors are defined as the following:

  * - DCIS: Estrogen receptor (ER) positive (>= 60%)
  * Invasive breast cancer:

    * Oncotype DX =< 25 (if performed) OR
    * If Oncotype DX is not performed an Allred score of 7 or 8. The following combinations of proportion of ER positive cells and staining intensity are allowed:

      * ER positive (34-66% of cells) and staining intensity is strong (Allred 7)
      * ER positive (>= 67% of cells) and staining intensity is intermediate (Allred 7)
      * ER positive (>= 67% of cells) and staining intensity is strong (Allred 8)
* Tissue from core biopsy or resection must be HER2 negative by current American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines
* Patients must have undergone breast conserving surgery with resulting negative surgical margins (no tumor on ink). Re-excision for negative margins is allowed. Patients with pathologically involved surgical margins are excluded
* Patients must have pathologic Tis or T1 disease
* Patients with invasive breast cancer, including patients with microinvasion, must have undergone surgical staging of the axilla (sentinel lymph node biopsy or axillary lymph node dissection) and have pathologically confirmed uninvolved lymph nodes. All lymph nodes must be pathologically negative (pN0[i-]). pN0(i+), pN1mic, pN1-pN3 axillary lymph nodes are not allowed Although an axillary lymph node dissection is not anticipated for low-risk ER positive breast cancers, axillary lymph node dissection is permissible
* Patient must have physician-reported "excellent" or "good" cosmesis post-lumpectomy and prior to radiation therapy based on the 4-point Global Cosmetic Score
* Women of childbearing potential (WOCBP): Negative urine or serum pregnancy test.

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females of childbearing potential* to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 1 month after the last dose of protocol therapy

  * Childbearing potential is defined as not being surgically sterilized or have not been free from menses for > 1 year

Exclusion Criteria:

* Any prior treatment with radiation therapy, anti-endocrine/hormone therapy, chemotherapy or biologic therapy for the currently diagnosed breast cancer PRIOR to surgical resection
* Prior radiation to the region of the involved breast that in the opinion of the investigator would preclude partial breast irradiation
* Clinically significant uncontrolled illness
* Diagnosis of Paget's disease of the nipple
* Other prior or active malignancy. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Pregnant or breastfeeding
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-09-29 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of women that rate the cosmetic appearance of the breast as acceptable ("excellent" or "good") | At 1 year post accelerated partial breast irradiation once daily (APBI QD)
  Measured by the 4-point Global Cosmetic Score (GCS). The exact test will be used to test the hypothesis that the rate of cosmesis is >= 90% versus the null hypothesis that cosmesis is 74% or lower, at the 5% significance level.

SECONDARY OUTCOMES:
Cosmetic outcome by the patient post-APBI QD | Over time at baseline, day 5, 1 month, 6 months, 1 year, 2 years and 3 years
  Measured by the GCS. Will be summarized and the percent and 95% confidence limits of the estimate will be calculated. Will also examine at cosmesis scores over time using analysis of variance (ANOVA).
Cosmetic outcome assessed by the physician post-APBI QD | At 1 year
  Measured by the GCS. Will explore also examine change in scores over time using ANOVA. Appropriate graphical methods will be used for visualization. Association between the assessment rating of cosmetic outcome based on photographic image by medical doctor (MD) and blinded reviewers will be calculated at each time point using Pearson's product-moment correlation coefficient.
Cosmetic outcome assessed by the physician post-APBI QD | Over time at baseline, day 5, 1 month, 6 months 1 year, 2 years and 3 years
  Measured by the GCS. Will explore also examine change in scores over time using ANOVA. Association between the assessment rating of cosmetic outcome based on photographic image by MD and blinded reviewers will be calculated at each time point using Pearson's product-moment correlation coefficient.
Incidence of adverse events-patients reported | Up to 3 years post-APBI
  Scored by the Patient-Reported Outcome Common Terminology Criteria for Adverse Events (CTCAE). Will be summarized using standard methods.
Incidence of adverse events-treatment team reported | Up to 3 years post-APBI
  As scored by the treatment team using CTCAE version 5.0. Will be summarized using standard methods.
In-breast recurrence | Up to 5 years post-APBI QD
  The Kaplan-Meier method will be used along with 95% confidence intervals.
Regional recurrence | Up to 5 years post-APBI QD
  The Kaplan-Meier method will be used along with 95% confidence intervals.
Distant metastases | Up to 5 years post-APBI QD
  The Kaplan-Meier method will be used along with 95% confidence intervals.
Disease-free survival | Up to 5 years post-APBI QD
  The Kaplan-Meier method will be used along with 95% confidence intervals.
Overall survival | Up to 5 years post-APBI QD
  The Kaplan-Meier method will be used along with 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Jose G Bazan, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States